CLINICAL TRIAL: NCT06653023
Title: A Clinical Study on the Safety and Efficacy of Universal CAR-T Cells (REVO-UWD-03) for Advanced Hepatocellular Carcinoma &Amp; Lung Cancer
Brief Title: Universal CAR-T Cells (REVO-UWD-03) for Advanced Hepatocellular Carcinoma and Lung Cancer
Acronym: Wondercel-UWD3
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wondercel Biotech (ShenZhen) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-REVO-UWD-03
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HCC - Hepatocellular Carcinoma; NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: Universal CAR-T cells; Allogeneic CAR-T therapy; Wondercel REVO U-CAR platform
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose injection of REVO-UWD-03 (Experimental): Dose escalation will be performed for the single dose injection of REVO-UWD-03 for treating HCC and NSCLC
  Interventions: Biological: Universal CAR-T cells injection for treating HCC and NSCLC; Drug: MMF Immunosuppression

INTERVENTIONS:
Biological: Universal CAR-T cells injection for treating HCC and NSCLC — Eligible participants will undergo FC lymphodepleting chemotherapy preconditioning after signing an informed consent form, followed by a one-time injection of one dose of universal REVO-UWD-03 CAR-T cells
  Other Names: REVO-UWD-03
Drug: MMF Immunosuppression — One day after the completion of fludarabine preconditioning (D-2), initiate oral mycophenolate sodium at a dose of 1440 mg twice daily (BID) for 15 consecutive days, or extend the duration appropriately based on CAR-T cell expansion status (discontinuation may occur at the end of CAR-T cell expansion or on the day of patient discharge). The maximum duration of administration must not exceed 30 days.

SUMMARY:
This is an investigator initiated trial to assess the efficacy and safety of a GPC3-targeting CAR-T therapy (REVO-UWD-03) in the HCC and Lung Cancer. It also aims to explore the feasibility of using a novel universal CAR-T cell platform.

DETAILED DESCRIPTION:
The study will use T cells from healthy donors, modified using a novel universal CAR-T technology, to treat HCC and Lung Cancer patients. The antigen-binding site of the CAR molecule recognizes GPC3 as the target.

The main questions it aims to answer are: • What is the maximum tolerated dose (MTD) of GPC3-CAR-T therapy in universal CAR-T cell treatments? • What are the dose-limiting toxicities (DLT) and treatment-emergent adverse events (TEAE)? • What is the treatment efficacy, as measured by objective response rate (ORR) and progression-free survival (PFS)? Researchers will assess whether the universal CAR-T cells have good safety and efficacy in treating HCC or Lung cancer, while improving accessibility and lowering treatment costs. Participants will: • Receive universal GPC3-CAR-T cells through a 3+3 dose escalation scheme. • Undergo chemotherapy conditioning before CAR-T infusion. • Be monitored for adverse events, immune response, and disease progression.

The study will collect data on both short-term outcomes (within the first few months post-treatment) and long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years and ≤75 years;
2. Patients with histologically or cytologically confirmed, unresectable locally advanced or metastatic epithelial-origin hepatocellular carcinoma (HCC) who have failed standard therapy, or for whom no standard therapy is available, or who are unsuitable for standard therapy at this stage;

(1) Barcelona Clinic Liver Cancer (BCLC) stage B (not amenable to hepatic surgery and/or other local therapies, or disease progression after local therapy) or stage C; (2) Or China Liver Cancer (CNLC) stage IIb or III (not amenable to hepatic surgery and/or other local therapies, or disease progression after local therapy); 3. Immunohistochemistry (IHC) evaluation showing GPC3 expression ≥1+ in ≥50% of the tumor lesion area (randomly select at least 5 fields of view from tumor regions for evaluation; at least 5 unstained slides must be provided for assessment); 4. At least one measurable lesion: The measurable lesion must not have received prior radiotherapy, interventional therapy, or other local treatments (lesions in previously treated fields may be selected as target lesions if confirmed to have progressed); 5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; 6. Expected survival ≥90 days; 7. Adequate major organ function, meeting the following criteria:

1. Hematology: Absolute neutrophil count ≥1.5 × 10⁹/L; platelets ≥80 × 10⁹/L; hemoglobin ≥9.0 g/dL;
2. Liver function: Total bilirubin ≤5 × upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 × ULN;
3. Renal function: Serum creatinine ≤5 × ULN or estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73 m²;
4. Coagulation: Prothrombin time (PT) prolongation ≤4 seconds;
5. Cardiac function: Left ventricular ejection fraction (LVEF) >50%; 8. No hemorrhagic disorders or coagulopathy; 9. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment, and agree to use appropriate contraception from enrollment through 8 weeks after the last CAR-T administration (women who have undergone sterilization or been postmenopausal for at least 2 years are considered not of childbearing potential); 10. Voluntary participation in the study, signed informed consent, good compliance, and willingness to complete follow-up.

Exclusion Criteria

1. Pregnant or breastfeeding women;
2. Received chemotherapy, targeted therapy, other investigational drugs, or monoclonal antibody therapy within 14 days prior to cell collection;
3. Participated in another drug clinical trial within 4 weeks prior to study initiation;
4. Any of the following cardiovascular diseases or cardiovascular risk factors:

(1) LVEF <50%; (2) New York Heart Association (NYHA) Class III or IV; (3) History of myocarditis, cardiomyopathy, or myocardial infarction within 6 months prior to enrollment (unless cardiac function has recovered as assessed by the investigator); (4) Uncontrolled arrhythmias (e.g., atrial fibrillation, ventricular tachycardia) or requiring long-term antiarrhythmic therapy; (5) QTcF interval >480 ms on screening ECG; (6) Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg); (7) History of ischemic or hemorrhagic stroke (unless stable for >6 months with no sequelae); (8) Uncontrolled intracranial lesions (e.g., brain tumors, aneurysms); (9) History of deep vein thrombosis (DVT) or pulmonary embolism (PE) (unless treated with anticoagulation for ≥6 months and stable); (10) Significantly elevated troponin or BNP/NT-proBNP levels suggestive of potential cardiac injury or dysfunction; 5. Non-healing wounds or fractures for a prolonged period; 6. History of substance abuse (including psychiatric drugs) that cannot be discontinued, or history of psychiatric disorders; 7. Uncontrolled or active fungal, bacterial, viral, or other infections; 8. Active or documented gastrointestinal bleeding within 6 months (e.g., esophageal varices or ulcer bleeding); 9. Prior antitumor treatment-related toxicities not recovered to ≤Grade 1 (or to the level specified in inclusion/exclusion criteria); 10. Known HIV infection; known active syphilis infection; or active hepatitis B (HBsAg positive and HBV-DNA ≥500 IU/mL or above the lower limit of detection, whichever is higher) or hepatitis C virus (anti-HCV positive and HCV-RNA above the lower limit of detection) infection; 11. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage despite appropriate intervention; 12. Severe allergic reaction history to key study drugs (including fludarabine, cyclophosphamide, mycophenolate sodium, tocilizumab, and anti-infective agents used during preconditioning); 13. Active autoimmune disease requiring systemic treatment within 2 years (including but not limited to autoimmune hepatitis, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, etc.); physiologic corticosteroid replacement therapy (e.g., thyroxine, insulin, or corticosteroids for adrenal or pituitary insufficiency) is not considered systemic treatment; 14. Female subjects unwilling to use contraception from informed consent signing through 6 months after CAR-T cell infusion; 15. Patients with meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, or active/symptomatic central nervous system (CNS) metastases not treated locally; 16. History of interstitial lung disease (ILD) or non-infectious pneumonitis requiring steroid treatment; 17. Clinically significant pulmonary impairment due to underlying lung disease, including but not limited to any baseline pulmonary disease (e.g., pulmonary embolism within 3 months prior to enrollment, severe asthma, severe chronic obstructive pulmonary disease), or any autoimmune, connective tissue, or inflammatory disease that may involve the lungs (e.g., rheumatoid arthritis, sarcoidosis), or prior pneumonectomy; 18. Any condition that, in the investigator's opinion, interferes with drug evaluation, participant safety, or study outcomes, or any other condition deemed unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-10-20 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within the first month post-infusion
  The highest dose of universal GPC3-CAR-T cells that can be administered without causing unacceptable side effects, measured during the dose escalation phase.
Dose-Limiting Toxicities (DLT) | Within the first month post-infusion.
  The incidence of treatment-related toxicities that prevent further dose escalation.
Treatment-Emergent Adverse Events (TEAE) | From the administration of UWD-03 CAR-T cells through six months post-infusion
  The frequency and severity of adverse events that arise following the administration of universal GPC3-CAR-T cells.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Measured at 3 and 6 months after treatment.
  The proportion of patients with a measurable reduction in tumor size (complete or partial response) following universal GPC3-CAR-T therapy.
Progression-Free Survival (PFS) | From the start of treatment up to 5 years.
  The length of time during and after treatment that the patient lives without disease progression.
Overall Survival (OS) | From the start of treatment up to 5 years.
  The duration from the start of treatment to the time of death from any cause.
Duration of Response (DOR) | From the administration of UWD-03 CAR-T cells to a maximum follow-up period of five years.
  The time from initial tumor response (CR or PR) to disease progression or relapse.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jiangsu Cancer Hospital, Nanjing

IPD SHARING:
Plan to Share IPD: No